CLINICAL TRIAL: NCT02575469
Title: Exercise Capacity in Diseases and Health
Status: Not yet recruiting | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Prof. Avraham Lorber, Head of pediatric cardiology institute, Ruth children hospital, Rambam Health Care Campus
Other Study IDs: 0323-14- RMB-CTIL
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Exercise Capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Exercise capacity is a key factor to evaluate and treat patients in different diseases (e.g. ischemic heart disease, chronic obstructive pulmonary disease, cystic fibrosis). The best way to measure exercise capacity is to perform a cardiopulmonary exercise testing. Normal/reference values in health and disease relate to specific population and subpopulations. The population in Israel is unique in its diversity.

Objectives: Data collection of exercise capacity assessment in health and illness in the northern of Israel for future local database.

Population: 500 Patients evaluated routinely in the exercise lab (pediatric cardiology institute) and healthy volunteers evaluated as controls.

Study design: Prospective observational study. Participants will answer a health related questioner, undergo a physical examination, perform a cardiopulmonary exercise test on a treadmill or a cycle ergometer.

DETAILED DESCRIPTION:
Exercise capacity is a key factor to evaluate and treat patients in different diseases (e.g. ischemic heart disease, chronic obstructive pulmonary disease, cystic fibrosis). The best way to measure exercise capacity is to perform a cardiopulmonary exercise testing. Normal/reference values in health and disease relate to specific population and subpopulations. The population in Israel is unique in its diversity.

Objectives: Data collection of exercise capacity assessment in health and illness in the northern of Israel for future local database.

Population: 500 Patients evaluated routinely in the exercise lab (pediatric cardiology institute) and healthy volunteers evaluated as controls.

Study design: Prospective observational study. Participants will answer a health related questioner, undergo a physical examination, perform a cardiopulmonary exercise test on a treadmill or a cycle ergometer .

ELIGIBILITY:
Inclusion Criteria:

* Ability to complete full exercise evaluation (including cardiopulmonary exercise testing).

Exclusion Criteria:

* Acute illness on visit day.
* for healthy volunteers: chronic disease or use of medications.
* Professional athletes.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 500 Patients evaluated routinely in the exercise lab (pediatric cardiology institute) and healthy volunteers evaluated as controls.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2035-10-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
VO2 (oxygen consumption) | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- RAMBAM health care center, Haifa, Israel